CLINICAL TRIAL: NCT02274207
Title: Phase IV Study of Antibacterial Effect on Silver Dressing of NPWT
Brief Title: Comparative Study of Antibacterial Effect on Silver Dressing of Negative Pressure Wound
Acronym: NPWT-silver
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Woojin Choi, Orthopedics, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SS-14-NPWT; CGBIOW1404 (Other Grant/Funding Number: CGBIO CO., LTD.)
Record Dates: First submitted 2014-09-02; First posted 2014-10-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes Mellitus
Keywords: Silver dressing; NPWT; DMF; foot
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- silver dressing (Experimental): Frequency and duration : 1 change/1day or according to statue of patient Dosage : 1 ea
  Interventions: Device: NPWT application
- non-silver dressing (Active Comparator): Frequency and duration : 1 change/1day or according to statue of patient Dosage : 1 ea
  Interventions: Device: NPWT application

INTERVENTIONS:
Device: NPWT application — NPWT mode is cyclic mode : -125~-50 mmHg

SUMMARY:
The purpose of this study is to test therapeutic benefits of silver dressing compared with non-silver dressing in NPWT(Negative pressure wound therapy). Silver dressing may antibacterial effect on infected diabetes mellitus foot.

DETAILED DESCRIPTION:
Investigator will recruit sixty patients. Participant will be randomly assigned to one of two groups. One is using silver dressing group in NPWT, another is using non-silver dressing group in NPWT. Participant will visit in screening day, NPWT apply day and F/u day for 4 months. Investigators will conduct to check the wound base, Lab, wound culture.

ELIGIBILITY:
Inclusion Criteria:

* The patient above 20 years and has type I, II of diabetes mellitus foot ulcer
* Infected ulcer has one of below.

  1. clinically infection symptom in ulcer area : warmth, erythema, tenderness/swelling

     * induration, purulent discharge etc.
  2. Confirmed case of bacteria in wound culture.
  3. Conformed case of abnormal range of erythrocyte sedimentation rate (ESR)/C-reactive protein(CRP) level in lab.
* Has to be applied NPWT because suture is impossible in ulcer area.
* The patient voluntary agreed to this protocol.
* In the opinion of investigator, It is suitable to participate in this study.

Exclusion Criteria:

* Infection in bone so patient need amputation
* Female with childbearing, lactating or not agree to prevent pregnancy.
* Has Sepsis, Osteomyelitis
* Has Connective tissue disease of disturbance of healing of wound Ex) Rheumarthritis,systemic lupus erythematosus(SEL), myalgia.
* The patient to diagnosis of Sickle sell disease or Charcot's joint.
* The patient stability treated chronic wasting disease.
* Malignant tumor or history of malignant disease. (Not diagnosis of complete recovery.)
* The patient treated chemotherapy, radiation therapy, immune-suppressants therapy,adrenocortical hormones therapy.
* Although necrosis tissue is removed, the target ulcer did not heal because of gangrenous, necrosis tissue or purulent pyorrhea.
* Has ulcer with cardiac arrhythmia thrombus, venous insufficiency, diabetic necrobiosis lipoidic.
* In case of using prohibited concomitant medications during study.

  a. Oral system steroid b. Immune-suppressive drug c. Unfractionated heparin infusion d. improper drugs in the opinion of investigator.
* Hypersensitivity with applicators. (NPWT, Silver)
* The patient participated in other clinical trials within 30 days
* In the opinion of investigator, the patient is not suitable to participate in this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-05 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Days to patient discharge | up to 4 weeks
  -Examine the days from applied medical device to discharge.

SECONDARY OUTCOMES:
Days to infection clearance in wound culture results | 4 months (at least once a week for 4 weeks / After dischage, every participant visit day(for 3 months))
  * Compare screening culture test with every visit culture test
  * Examine days to infection clearance(point to show bacteria minus level in culture test)
Complete infection clear rate in wound culture results | up to 4 months
  * Compare screening culture test with every visit culture test
  * Examine total complete infection clear rate in each groups. (point to show bacteria minus level in culture test)
Days to complete wound closure | 4 months (at least once a week for 4 weeks / After dischage, every participant visit day(for 3 months))
  -Examine days from applied medical device to wound closure day
Wound closure rate | up to 4 months
  * Examine total wound closure rate in each groups.
  * Wound closure: definition: skin graft, epithelized skin or simple suture et. al.
Elevation of wound evaluations grade | 4 months (at least once a week for 4 weeks / After dischage, every participant visit day(for 3 months))
  * Examine the rate of wound size, wound depth (4 category),granulation tissue grade (5 step),Infection symptom(4 grade)
  * Present wound size, infection grade, depth category, granulation tissue grade at every patient visit and examine elevation of wound evaluations compared with baseline.
Days of NPWT application period | up to 8 weeks
  -Examine the period of NPWT application
Number of surgical debridement after NPWT | up to 8 weeks
  -Examine the number of debridement during applied NPWT
Lab - deviation of level | up to 4 months
  * Compared baseline lab level
  * Examine related infection sign level (white blood cell,monocytes,C-reactive protein)
  * Finding adverse deviation level through the lab level
Rate of adverse event | up to 4 months (if adverse event appeared, Investigator follow until the disappearance of the symptom
  -Examine adverse event every visit

CONTACTS AND LOCATIONS:
Overall Officials: WooJin Choi, MD, Principal Investigator — Korea: Severance hospital
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea